CLINICAL TRIAL: NCT04306081
Title: Effect of Evolocumab in Functional Status and LDL Oxidation of Patients With Peripheral Arterial Disease (Evol-PAD)
Brief Title: Effect of Evolocumab in Functional Status and LDL Oxidation of Patients With Peripheral Arterial Disease
Acronym: Evol-PAD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Leonardo Clavijo (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor-Investigator, Leonardo Clavijo, Associated Professor Cardiology, USC. Director Vascular Medicine and Peripheral Interventions Program Director, Interventional Cardiology Fellowship, University of Southern California, University of Southern California
Organization: University of Southern California (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20167764; HS-16-00965 (Other: University of Southern California)
Record Dates: First submitted 2020-02-21; First posted 2020-03-12 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Peripheral Arterial Disease
Keywords: PAD; Hyperlipidemia; Claudication
MeSH Terms: conditions — Peripheral Arterial Disease; Hyperlipidemias; Intermittent Claudication | interventions — evolocumab

STUDY DESIGN:
Intervention Model Description: This is a double-blinded, prospective, randomized, placebo-controlled study.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study subjects will be randomized, to receive either evolocumab or placebo. Each participant will have equal chance of receiving evolocumab or placebo. The study participant, the care provider and the investigator will not know to which study arm the participant was assigned.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Arm (Experimental): 43 Patients with lower extremities Peripheral Arterial Disease on maximum statin therapy will receive in addition a monthly dose of evolocumab 420 mg via subcutaneous injections for 6 months.
  Interventions: Drug: Evolocumab 140 mg/mL Subcutaneous Injection 1 milliliter (mL) pre-filled injector Pen x 3 for a monthly dose of 420 mg for 6 months.
- Control Arm (Placebo Comparator): 43 Patients with lower extremities Peripheral Arterial Disease on maximum statin therapy will receive in addition a monthly dose of placebo via subcutaneous injections for 6 months.
  Interventions: Other: Placebo 1milliliter (mL) Subcutaneous Injection pre-filled injector Pen x 3 monthly for 6 months.

INTERVENTIONS:
Drug: Evolocumab 140 mg/mL Subcutaneous Injection 1 milliliter (mL) pre-filled injector Pen x 3 for a monthly dose of 420 mg for 6 months. — The study subjects randomized to the treatment study arm will receive monthly subcutaneous injections of evolocumab 420 mg in the abdomen, thigh or upper arm. The study drug (evolocumab) prefilled injector pens are provided by Amgen
  Other Names: Repatha
  Arms: Treatment Arm
Other: Placebo 1milliliter (mL) Subcutaneous Injection pre-filled injector Pen x 3 monthly for 6 months. — The study subjects randomized to the treatment study arm will receive monthly subcutaneous injections of Placebo in the abdomen, thigh or upper arm. The Placebo prefilled injector pens are provided by Amgen
  Other Names: Control
  Arms: Control Arm

SUMMARY:
Peripheral arterial disease (PAD) is a manifestation of systemic atherosclerotic cardiovascular disease (ASCVD) and is associated with increase cardiovascular risk. PAD impairs quality of life due to symptoms of claudication, pain at rest or risk of limb loss.

All major societies recognize the importance of LDL reduction in patients with PAD.

Statin therapy improves cardiovascular end-points in patients with PAD and have been shown to improve symptoms of lower extremity intermittent claudication (pain free walking time), 6-minute walking time, ankle-brachial index (ABI), and endothelial function, while decreasing markers of atherosclerosis.

This study aims to demonstrate that in patients with PAD on stable maximal tolerated lipid lowering regimen with a statin, further reduction of LDL with the pro protein converts subtilisin/kexin type 9 (PCSK-9) inhibitor Evolocumab, improves functional status (pain free walking time in particular, but also maximal walking time), lower extremity arterial perfusion and endothelial function (brachial endothelial reactivity).

DETAILED DESCRIPTION:
This is a double-blinded, prospective, randomized, study in eighty-six subjects with clinical ASCVD with PAD on background treatment with maximal tolerated dose of a statin. Subjects will be assessed based on their medical history and physical examination. Eligible subjects must meet all inclusion criteria and none of the exclusion criteria (listed below). There will be a treatment group and a placebo group, each with equal number of participants (n=43 patients in each group). After consent and enrollment, subjects will have a venous blood sample drawn to perform serum circulating biomarkers of oxidative stress as oxidized low density lipoprotein (oxLDL), oxidized glutathione : reduced glutathione (GSH:GSSG) and soluble CD36 (sCD36). We will then perform: functional walking measurements, pain free walking time (PFWT), and (maximal walking time (MWT), lower extremity arterial perfusion assessment (rest ABI/TBI, post-exercise ABI and bilateral TcPO2), and brachial endothelial function testing (after hyperemia). Subjects will receive monthly subcutaneous injections of Evolocumab 420 mg or placebo injection. The study participants will be seen at three months and six months for follow up and a final assessment at 26 +/-2 weeks, all tests will be repeated for comparison from baseline and/or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent.
* Age ≥40 to ≤85 years of age at the time of consent.
* Diagnosis of ASCVD with peripheral arterial disease, Rutherford class I-VI at the time of diagnosis, confirmed by ABI≤0.9 at rest or ABI≤0.8 after exercise, angiography, duplex ultrasound or history of lower extremity surgical or endovascular revascularization.
* At least 1 months from last intervention, including surgery or endovascular procedures.
* Stable on maximal tolerated doses of a lipid-lowering regimen for at least 4 weeks.
* Most recent fasting LDL-C ≥55 mg/dL or non-HDL-C ≥80 mg/dL.

Exclusion Criteria:

* Subjects with active, non-healed wounds.
* Subjects with anticipated need of cardiac or surgical revascularization procedures.
* Subjects with chronic inflammatory conditions or requiring chronic systemic corticosteroids.
* New York Heart Association (NYHA) class III or IV heart failure, or known left ventricular ejection fraction <30%.
* Uncontrolled arrhythmia.
* Uncontrolled hypertension with systolic BP>180 mmHg or diastolic >100 mmHg.
* Untreated thyroid disease.
* Severe chronic renal disease with estimated glomerular filtration rate (eGFR) <20 mL/min.
* Liver disease with aspartame aminotransferase (AST) or alanine aminotransferase (ALT) ≥3 times the upper limit of normal.
* Status post-organ transplant.
* Pregnant and breastfeeding women
* Fertile age female not on appropriate birth control.
* Clinically significant disease that, in the opinion of the Principal Investigator, is likely to require surgery or immunotherapy that may interfere with the completion of the study.
* Active cancer or life expectancy of less than two years.
* Chronic anticoagulation or hypercoagulability disorder.
* Atrial fibrillation with a CHADS-VASc Score ≥2 or any clinical condition which, in the opinion of the Principal Investigator increases the risk of cerebrovascular events.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2017-12-14 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2021-03-30 (Estimated)

PRIMARY OUTCOMES:
Evolocumab effect in pain free walking time (PFWT) in patients with PAD | six months
  To evaluate change in pain free walking time (PFWT) in patients with PAD at baseline and after six months of therapy with Evolocumab.
  PFWT will be measured in minutes, using a graded treadmill Gardner protocol with a constant speed of 2 miles per hour, increasing by 2% grade every 2 minutes.

SECONDARY OUTCOMES:
Evolocumab effect in maximal walking time (MWT) in patients with PAD | six months
  To evaluate changes in maximal walking time (MWT) in patients with PAD at baseline and after six months of therapy with Evolocumab.
  MWT will be measured in minutes, using a graded treadmill Gardner protocol with a constant speed of 2 miles per hour, increasing by 2% grade every 2 minutes.

OTHER OUTCOMES:
Evolocumab effect in lower extremity arterial perfusion in ankle-brachial indices (ABI). | six months
  To evaluate changes in lower extremity arterial perfusion in patients with PAD at baseline and after 6 month therapy with evolocumab, measured by systolic pressure rate changes in ankle-brachial indices (ABI).
  The rest ABI will be calculated by the dorsalis pedis and posterior tibialis arteries highest systolic pressure value (in mmHg) of each foot divided by the brachial artery highest systolic pressure (in mmHg) of both arms.
Evolocumab effect in lower extremity arterial perfusion pressure in post-exercise ankle-brachial indices. | six months
  To evaluate changes in lower extremity arterial perfusion in patients with PAD at baseline and after 6 month therapy with evolocumab, measured by systolic pressure rate changes in post-exercise ankle-brachial indices (ABI).
  The post-exercise ABI will be calculated by the dorsalis pedis and posterior tibialis arteries highest systolic pressure value (in mmHg) of each foot divided by the brachial artery highest systolic pressure (in mmHg) of both arms and assessed by using a standardized treadmill walking protocol at a 2% progressive grade every 2 minutes and 2 miles per hour until symptoms force the subject to stop.
Evolocumab effect in lower extremity arterial perfusion pressure in Toe-Brachial pressure indices. | six months
  To evaluate changes in lower extremity arterial perfusion in patients with PAD at baseline and after 6 month therapy with evolocumab, measured by systolic pressure rate changes toe-brachial indices (TBI).
  The TBI will be determined by the great toe pressure value (in mmHg) of each foot divided by the brachial artery highest systolic pressure (in mmHg) of both arms.
Evolocumab effect in lower extremity arterial perfusion in transcutaneous oxygen changes. | six months
  To evaluate lower extremity arterial perfusion determined by changes in transcutaneous oxygen tension in the skin (in tcpo2 mmHg) at baseline and after 6 month therapy with evolocumab in patients with PAD.
  Transcutaneous oxygen will be performed by placing electrodes on the skin at different levels of each leg, foot and chest for reference.
Evolocumab effect in brachial endothelial function by changes in Flow Mediated Dilation (FMD). | six months
  To evaluate changes in brachial endothelial function FMD determined by brachial artery diameter in response to shear stress of both arms in patients with PAD at baseline and after six months of therapy with Evolocumab compared with placebo.
  The FMD will be measured as the percentage (%) change in brachial artery diameter from baseline in response to the increase flow achieved after the inflation of a pneumatic cuff to supra-systolic pressure for 5 minutes.
  The ultrasound brachial images will be acquired using a LOGIQ eR7 ultrasound and a 12-L-RS linear array transducer and the images will be analyzed by the QUIPU automated cardiovascular suite, FMD studio software.
Evolocumab effect in serum circulating biomarker oxidative LDL | six months
  To evaluate changes on LDL oxidation by measuring oxidized LDL levels (oxLDL), performed using a sandwich ELISA method in patients with PAD at baseline and after six months of therapy with Evolocumab.
Evolocumab effect in serum circulating biomarker soluble CD36 (sCD36). | six months
  To evaluate changes on human soluble CD36 levels at baseline and after 6 month therapy with evolocumab in patients with PAD by using a quantitative sandwich ELISA format.

CONTACTS AND LOCATIONS:
Overall Officials: Leonardo Clavijo, MD, PhD, Principal Investigator — University of Southern California
Locations (1):
- University of Southern California, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No